CLINICAL TRIAL: NCT04910958
Title: Impact of COVID-19 Pandemic on Early Spontaneous Abortions and Early Termination of Pregnancy
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0199-20-HYMC
Record Dates: First submitted 2021-06-01; First posted 2021-06-02 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Termination of Pregnancy; Covid19; Pregnancy Loss
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To see the impact the COVID-19 pandemic has had on early spontaneous abortions and early termination of pregnancy in the first trimester

DETAILED DESCRIPTION:
To date, the research has focused on the complications of SARS-CoV-2 in pregnant women. There is no research in the literature that has compared the rates and behavior of miscarriage during the time of the COVID-19 pandemic to before the time of the pandemic. As described in the literature, there is an established connection between COVID-19 and stress, anxiety, and depression. There is also an established connection between stress, anxiety, and depression and rates of miscarriage. The investigators hereby wish to analyze the effect of the COVID-19 pandemic on miscarriages.

In this study, The investigators will analyze the number of early missed abortions and number of termination of pregnancies in the first trimester before and during the COVID-19 pandemic. The investigators will also analyze the time interval between diagnosis of missed abortion and attendance to E.R in missed abortions during the COVID-19 pandemic. In addition, The investigators will be comparing the reasons for termination of pregnancy during this time, as well as analyzing age, religion, and demographic variables during the COVID-19 pandemic compared to years prior.

ELIGIBILITY:
Inclusion Criteria:

* All women attending for early missed abortion or termination of pregnancy receiving treatment between March 11th - November 30th during the years 2017-2020 Gestational age until 12 weeks 6 days (1st trimester only)

Exclusion Criteria:

* Incomplete and complete abortions
* Gestational age >13 weeks

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Females only
Study Population: All women attending for early missed abortion or termination of pregnancy receiving treatment between March 11th - November 30th during the years 2017-2020 Gestational age until 12 weeks 6 days (1st trimester only)
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Number of early missed abortions | Two years
  Number of early missed abortions in the first trimester in COVID19 time compared to years prior
Number of termination of pregnancies | Two years
  Number of termination of pregnancies in the first trimester in COVID19 time compared to years prior

SECONDARY OUTCOMES:
Time between discovery and attendance | 1 year
  Time between discovery and attendance in missed abortions during COVID19 time compared to years prior
Comparison of reasons for termination | 1 year
  Comparison of reasons for termination of pregnancy during COVID19 time compared to years prior
Comparison of Age/Religion/Demographic variables | 1 year
  Comparison of Age/Religion/Demographic variables of termination of pregnancy during COVID19 time compared to years prior

CONTACTS AND LOCATIONS:
Overall Officials: Omer Mor, MD, Principal Investigator — omer.moore@gmail.com
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel